CLINICAL TRIAL: NCT02067663
Title: Comparison of the Levonorgestrel IUD and the Copper IUD Placed in the Immediate Postplacental Period: A Prospective Cohort Study
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor
Other Study IDs: 13-3264
Record Dates: First submitted 2014-02-11; First posted 2014-02-20 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-06

CONDITIONS: Contraception
Keywords: Postplacental IUD placement; LNG-IUS
MeSH Terms: interventions — Levonorgestrel; Intrauterine Devices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Mirena Group: Women who have a postplacental Mirena IUD placed. (LNG-IUS)
  Interventions: Drug: Mirena
- Paragard Group: Women who have a postplacental Paragard IUD placed. (Copper IUD - T380A)
  Interventions: Device: Paragard

INTERVENTIONS:
Device: Paragard — The IUD will be placed as part of standard clinical care.
  Other Names: T380A IUD
  Groups: Paragard Group
Drug: Mirena — The IUD will be placed as part of standard clinical care.
  Other Names: LNG-IUS, IUD
  Groups: Mirena Group

SUMMARY:
The intrauterine device (IUD) is a safe, highly effective, long acting, and reversible form of contraception. The postpartum period is an important moment for contraceptive intervention; however there are many barriers to women obtaining birth control postpartum. The use of the IUD in the immediate postpartum setting offers many advantages and is considered safe, but the risk of expulsion appears to be higher than with interval insertion. Previous studies have shown the rate of expulsion of the copper IUD in the postplacental period to be in the range of 1-14% by 6-12 months, while the only study of the levonorgestrel IUD in the postplacental period documented a rate of expulsion of 24% by 12 months. While studies related to the copper IUD use ring forceps or the operator's hand for placement of the IUD, the only published study investigating immediate postplacental levonorgestrel IUD insertion utilized the manufacturer's inserter for IUD placement. The investigators therefore ask the question, is there a difference in expulsion rates between levonorgestrel and copper IUDs placed post-placentally when all providers undergo a standardized training, use a standardized insertion technique, and when patient level characteristics are controlled by randomization?

The investigators propose to perform a prospective cohort trial comparing the rates of expulsion for the levonorgestrel and the copper IUD by 3 months postpartum when placed in the uterus within 10 minutes of the delivery of the placenta, using a standardized technique (placement with a ring forceps or the operator's hand) after all providers undergo a formal didactic and skills training. The investigators hypothesis is that the levonorgestrel IUD has a higher rate of expulsion as compared to the copper IUD. Additional objectives include a comparison of the rates of complete IUD expulsion, partial IUD expulsion, unrecognized expulsions, complications, IUD continuation, pregnancy, and satisfaction. Additionally, the investigators will document the natural history of the location of the IUD within the uterus when placed in the immediate postpartum period, utilizing ultrasound at 24 hours, 6 weeks, and 3 months postpartum, to better understand the relationship between position of the IUD and subsequent expulsion.

ELIGIBILITY:
Inclusion Criteria:

* Women age ≥ 18
* Desire for immediate postpartum IUD or postpartum day #1 after a postplacental IUD placement
* English or Spanish speaking
* Willing to attend 2 follow-up visits

Exclusion Criteria:

* Multiple gestations
* Delivery prior to 35 weeks gestational age
* Allergy or sensitivity to any component of either IUD (including polyethylene, levonorgestrel or copper)
* Cesarean delivery
* Postpartum hemorrhage (estimated blood loss > 500 mL)
* Chorioamnionitis
* Abnormal uterine anatomy (including uterine anomaly or large fibroids)
* Treated for Chlamydia or Gonorrhea during pregnancy without a subsequent negative follow-up test
* Current cervical cancer or carcinoma in situ
* Current breast cancer
* Wilson's disease
* If enrolling postpartum after IUD has already been placed, women will be excluded if the provider used an insertion technique other than using the ring forceps or the operator's hand

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women interested in an immediate postpartum IUD, or those who recently had one placed, who are willing to be followed postpartum.
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2014-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Teal, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Winner B, Peipert JF, Zhao Q, Buckel C, Madden T, Allsworth JE, Secura GM. Effectiveness of long-acting reversible contraception. N Engl J Med. 2012 May 24;366(21):1998-2007. doi: 10.1056/NEJMoa1110855. PMID 22621627
- [Background] Thonneau PF, Almont T. Contraceptive efficacy of intrauterine devices. Am J Obstet Gynecol. 2008 Mar;198(3):248-53. doi: 10.1016/j.ajog.2007.10.787. Epub 2008 Jan 25. PMID 18221924
- [Background] ACOG Practice Bulletin No. 121: Long-acting reversible contraception: Implants and intrauterine devices. Obstet Gynecol. 2011 Jul;118(1):184-196. doi: 10.1097/AOG.0b013e318227f05e. No abstract available. PMID 21691183
- [Background] d'Arcangues C. Worldwide use of intrauterine devices for contraception. Contraception. 2007 Jun;75(6 Suppl):S2-7. doi: 10.1016/j.contraception.2006.12.024. Epub 2007 Apr 19. PMID 17531612
- [Background] Finer LB, Zolna MR. Unintended pregnancy in the United States: incidence and disparities, 2006. Contraception. 2011 Nov;84(5):478-85. doi: 10.1016/j.contraception.2011.07.013. Epub 2011 Aug 24. PMID 22018121
- [Background] Mosher WD, Jones J. Use of contraception in the United States: 1982-2008. Vital Health Stat 23. 2010 Aug;(29):1-44. PMID 20939159
- [Background] Allen RH, Goldberg AB, Grimes DA. Expanding access to intrauterine contraception. Am J Obstet Gynecol. 2009 Nov;201(5):456.e1-5. doi: 10.1016/j.ajog.2009.04.027. Epub 2009 Jun 13. PMID 19527902
- [Background] Jackson RA, Schwarz EB, Freedman L, Darney P. Advance supply of emergency contraception. effect on use and usual contraception--a randomized trial. Obstet Gynecol. 2003 Jul;102(1):8-16. doi: 10.1016/s0029-7844(03)00478-2. PMID 12850599
- [Background] Conde-Agudelo A, Rosas-Bermudez A, Kafury-Goeta AC. Birth spacing and risk of adverse perinatal outcomes: a meta-analysis. JAMA. 2006 Apr 19;295(15):1809-23. doi: 10.1001/jama.295.15.1809. PMID 16622143
- [Background] Zhu BP, Rolfs RT, Nangle BE, Horan JM. Effect of the interval between pregnancies on perinatal outcomes. N Engl J Med. 1999 Feb 25;340(8):589-94. doi: 10.1056/NEJM199902253400801. PMID 10029642
- [Background] Speroff L, Mishell DR Jr. The postpartum visit: it's time for a change in order to optimally initiate contraception. Contraception. 2008 Aug;78(2):90-8. doi: 10.1016/j.contraception.2008.04.005. Epub 2008 Jun 12. No abstract available. PMID 18672108
- [Background] Ogburn JA, Espey E, Stonehocker J. Barriers to intrauterine device insertion in postpartum women. Contraception. 2005 Dec;72(6):426-9. doi: 10.1016/j.contraception.2005.05.016. Epub 2005 Aug 9. PMID 16307964
- [Background] Grimes DA, Lopez LM, Schulz KF, Van Vliet HA, Stanwood NL. Immediate post-partum insertion of intrauterine devices. Cochrane Database Syst Rev. 2010 May 12;(5):CD003036. doi: 10.1002/14651858.CD003036.pub2. PMID 20464722
- [Background] Comparative multicentre trial of three IUDs inserted immediately following delivery of the placenta. Contraception. 1980 Jul;22(1):9-18. doi: 10.1016/0010-7824(80)90112-2. PMID 7418410
- [Background] Chi IC, Wilkens L, Rogers S. Expulsions in immediate postpartum insertions of Lippes Loop D and Copper T IUDs and their counterpart Delta devices--an epidemiological analysis. Contraception. 1985 Aug;32(2):119-34. doi: 10.1016/0010-7824(85)90101-5. PMID 3907964
- [Background] Celen S, Moroy P, Sucak A, Aktulay A, Danisman N. Clinical outcomes of early postplacental insertion of intrauterine contraceptive devices. Contraception. 2004 Apr;69(4):279-82. doi: 10.1016/j.contraception.2003.12.004. PMID 15033401
- [Background] Eroglu K, Akkuzu G, Vural G, Dilbaz B, Akin A, Taskin L, Haberal A. Comparison of efficacy and complications of IUD insertion in immediate postplacental/early postpartum period with interval period: 1 year follow-up. Contraception. 2006 Nov;74(5):376-81. doi: 10.1016/j.contraception.2006.07.003. Epub 2006 Sep 15. PMID 17046378
- [Background] Morrison C, Waszak C, Katz K, Diabate F, Mate EM. Clinical outcomes of two early postpartum IUD insertion programs in Africa. Contraception. 1996 Jan;53(1):17-21. doi: 10.1016/0010-7824(95)00254-5. PMID 8631184
- [Background] Xu JX, Rivera R, Dunson TR, Zhuang LQ, Yang XL, Ma GT, Chi IC. A comparative study of two techniques used in immediate postplacental insertion (IPPI) of the Copper T-380A IUD in Shanghai, People's Republic of China. Contraception. 1996 Jul;54(1):33-8. doi: 10.1016/0010-7824(96)00117-5. PMID 8804806
- [Background] Chen BA, Reeves MF, Hayes JL, Hohmann HL, Perriera LK, Creinin MD. Postplacental or delayed insertion of the levonorgestrel intrauterine device after vaginal delivery: a randomized controlled trial. Obstet Gynecol. 2010 Nov;116(5):1079-87. doi: 10.1097/AOG.0b013e3181f73fac. PMID 20966692
- [Background] Hayes JL, Cwiak C, Goedken P, Zieman M. A pilot clinical trial of ultrasound-guided postplacental insertion of a levonorgestrel intrauterine device. Contraception. 2007 Oct;76(4):292-6. doi: 10.1016/j.contraception.2007.06.003. Epub 2007 Aug 6. PMID 17900440
- [Background] Prescott GM, Matthews CM. Long-acting reversible contraception: a review in special populations. Pharmacotherapy. 2014 Jan;34(1):46-59. doi: 10.1002/phar.1358. Epub 2013 Oct 15. PMID 24130075
- [Background] Kapp N, Curtis KM. Intrauterine device insertion during the postpartum period: a systematic review. Contraception. 2009 Oct;80(4):327-36. doi: 10.1016/j.contraception.2009.03.024. Epub 2009 Aug 29. PMID 19751855
- [Background] Braaten KP, Benson CB, Maurer R, Goldberg AB. Malpositioned intrauterine contraceptive devices: risk factors, outcomes, and future pregnancies. Obstet Gynecol. 2011 Nov;118(5):1014-1020. doi: 10.1097/AOG.0b013e3182316308. PMID 22015868
- [Background] Inal MM, Ertopcu K, Ozelmas I. The evaluation of 318 intrauterine pregnancy cases with an intrauterine device. Eur J Contracept Reprod Health Care. 2005 Dec;10(4):266-71. doi: 10.1080/13625180500195340. PMID 16448955
- [Background] Sivin I, Stern J. Health during prolonged use of levonorgestrel 20 micrograms/d and the copper TCu 380Ag intrauterine contraceptive devices: a multicenter study. International Committee for Contraception Research (ICCR). Fertil Steril. 1994 Jan;61(1):70-7. doi: 10.1016/s0015-0282(16)56455-3. PMID 8293847
- [Background] Sivin I, el Mahgoub S, McCarthy T, Mishell DR Jr, Shoupe D, Alvarez F, Brache V, Jimenez E, Diaz J, Faundes A, et al. Long-term contraception with the levonorgestrel 20 mcg/day (LNg 20) and the copper T 380Ag intrauterine devices: a five-year randomized study. Contraception. 1990 Oct;42(4):361-78. doi: 10.1016/0010-7824(90)90046-x. PMID 2124179
- [Background] Andersson K, Odlind V, Rybo G. Levonorgestrel-releasing and copper-releasing (Nova T) IUDs during five years of use: a randomized comparative trial. Contraception. 1994 Jan;49(1):56-72. doi: 10.1016/0010-7824(94)90109-0. PMID 8137626
- [Background] Centers for Disease Control and Prevention (CDC). Update to CDC's U.S. Medical Eligibility Criteria for Contraceptive Use, 2010: revised recommendations for the use of contraceptive methods during the postpartum period. MMWR Morb Mortal Wkly Rep. 2011 Jul 8;60(26):878-83. PMID 21734635
- [Background] De la Cruz D, Cruz A, Arteaga M, Castillo L, Tovalin H. Blood copper levels in Mexican users of the T380A IUD. Contraception. 2005 Aug;72(2):122-5. doi: 10.1016/j.contraception.2005.02.009. PMID 16022851
- [Background] The TCu380A, TCu220C, multiload 250 and Nova T IUDS at 3,5 and 7 years of use--results from three randomized multicentre trials. World Health Organization. Special Programme of Research, Development and Research Training in Human Reproduction: Task Force on the Safety and Efficacy of Fertility Regulating Methods. Contraception. 1990 Aug;42(2):141-58. PMID 2085966
- [Background] Long-term reversible contraception. Twelve years of experience with the TCu380A and TCu220C. Contraception. 1997 Dec;56(6):341-52. PMID 9494767

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This prospective cohort trial was conducted at 2 affiliated teaching hospitals: University of Colorado Hospital (UCH) in Aurora, CO, and Denver Health Medical Center (DHMC) in Denver, CO.
Period: Overall Study
Arm/Group | Mirena Group | Paragard Group
Started | 68 | 55
Completed | 55 | 41
Not Completed | 13 | 14
Not completed — Lost to Follow-up | 13 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mirena Group | Paragard Group | Total
Number analyzed (Participants) | 68 | 55 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.2 (5.3) | 27.4 (5.4) | 26.72 (5.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 55 | 123
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 36 | 62
  Not Hispanic or Latino | 42 | 19 | 61
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 9 | 28
  White | 38 | 36 | 74
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 11 | 10 | 21
Region of Enrollment [Number; unit: participants]
  United States | 68 | 55 | 123

OUTCOME MEASURES:

1. Primary Outcome: IUD Expulsion Rate
Description: The primary outcome of the study is the total number of expulsions in the full 3 month study period. The provider will perform a speculum exam and transvaginal ultrasound. If expulsion has occurred, the participant will have an abdominal x-ray to confirm.
Time Frame: 3 months postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Mirena Group | Paragard Group
Number analyzed (Participants) | 55 | 41
Participants | 20 | 7

2. Secondary Outcome: Pregnancy
Description: A urine pregnancy test will be performed at the 6 week follow up visit if clinically indicated.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Mirena Group | Paragard Group
Number analyzed (Participants) | 56 | 45
Participants | 0 | 0

3. Secondary Outcome: Pregnancy
Description: A urine pregnancy test will be performed at the 3 month follow up visit if clinically indicated.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mirena Group | Paragard Group
Number analyzed (Participants) | 56 | 45
Participants | 0 | 0

4. Secondary Outcome: Complications
Description: A questionnaire will be administered to determine if the participant has had any complications since placement. Number of women reporting complications are reported.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mirena Group | Paragard Group
Number analyzed (Participants) | 55 | 41
Participants | 0 | 0

5. Secondary Outcome: Satisfaction
Description: A questionnaire will be administered to determine the participant's satisfaction level with the IUD. Satisfaction levels of >= 8 are reported by percent of participants.
Time Frame: 3 months
Measure: Number; unit: percent of participants
Arm/Group | Mirena Group | Paragard Group
Number analyzed (Participants) | 35 | 34
percent of participants | 91.4 | 94.2

6. Secondary Outcome: Intrauterine Device Expulsion (Day 1)
Description: Number of expulsions at Day 1. Position of the IUD within the uterus will be documented by ultrasound.
Time Frame: Day 1
Measure: Number; unit: participants
Arm/Group | Mirena Group | Paragard Group
Number analyzed (Participants) | 56 | 45
participants | 0 | 0

7. Secondary Outcome: Intrauterine Device Expulsion (6 Weeks)
Description: Number of expulsions. Position of the IUD within the uterus will be documented by ultrasound.
Time Frame: 6 weeks
Measure: Number; unit: participants
Arm/Group | Mirena Group | Paragard Group
Number analyzed (Participants) | 56 | 45
participants | 18 | 6

8. Secondary Outcome: Intrauterine Device Expulsion by 12 Weeks Postpartum
Description: Position of the IUD within the uterus will be documented by ultrasound.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Mirena Group | Paragard Group
Number analyzed (Participants) | 55 | 41
Participants | 21 | 8

ADVERSE EVENTS:
Time Frame: Adverse event information was collected from the time of consent until completion of participation (12 weeks).
Arm/Group | Mirena Group | Paragard Group
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/55
Other Adverse Events (participants affected / at risk) | 0/68 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No